CLINICAL TRIAL: NCT01097174
Title: A Multicenter Registry Study to Capture Data With Respect to CyPass Clinical Experience
Brief Title: CyPass Clinical Experience Study
Acronym: CyCLE
Status: Completed | Type: Observational
Sponsor: Transcend Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Other Study IDs: TMI-09-02
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2016-10

CONDITIONS: Open Angle Glaucoma (OAG)
Keywords: Glaucoma; Glaucoma device; Glaucoma surgery; Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CyPass Micro-stent: Patients in whom CyPass Micro-stent implantation was attempted.
  Interventions: Device: CyPass Micro-Stent

INTERVENTIONS:
Device: CyPass Micro-Stent — The CyPass Micro-Stent is a small tube with a through-lumen designed to redirect aqueous fluid from the front into the back of they eye.

SUMMARY:
This study is to evaluate the long-term safety, effectiveness and clinical experience of the CyPass Micro-Stent in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OAG
* IOP ≥ 21 mmHg and ≤ 31 mmHg (with or without ocular hypotensive medication)

Exclusion Criteria:

* Acute angle closure, narrow angle, uveitic or neovascular glaucoma
* Normal tension glaucoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2009-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative and postoperative adverse events | Day 0 - Year 3

SECONDARY OUTCOMES:
Intraocular pressure (IOP) reduction | 1 - 36 months postoperatively
Ocular hypotensive medication use | 1 - 36 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho (Sean) Ianchulev, MD, MPH, Study Director — Transcend Medical, Inc.
Locations (14):
- University Eye Clinic, Salzburg, Austria
- Specialized Hospital for Active Treatment of Ophthalmologic Diseases, Sofia, Bulgaria
- Germany (5):
  - Schlosspark-Klinik, Department of Ophthalmology, Berlin
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - AugenKlinik Cham, Cham
  - Klinik fur Augenheilkunde, Campus Lubeck, Lübeck
  - Klinik für Augenheilkunde, Dietrich-Bonhoeffer-Klinikum, Neubrandenburg
- Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazio, Catania, Italy
- Wojskowy Instytut Medyczny (Military Medical Institute), Warsaw, Poland
- Spain (5):
  - Institut Catala de Retina, Barcelona
  - Instituto de Microcirugia Ocular, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Ramón y Cajal University Hospital, Madrid
  - Hospital Universiatrio Miguel Servet, Zaragoza